CLINICAL TRIAL: NCT05885867
Title: The Effect of Dual Task Performance on the Activation and Walking Speed of the Prefrontal Cortex of the Elderly With Mild Cognitive Impairment During Straight and Curved Walking.
Brief Title: The Activation and Walking Speed of the Prefrontal Cortex of the Elderly Mild Cognitive Impairment During Dual Task.
Status: Completed | Type: Observational
Sponsor: Sahmyook University (Other)
Responsible Party: Principal Investigator, Yumin Lee, Physical Therapist, Sahmyook University
Other Study IDs: SYU 2023-02-013-002
Record Dates: First submitted 2023-04-26; First posted 2023-06-02 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Mild Cognitive Impairment; Dual Task
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Aging

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Seniors with mild cognitive impairment over 65 years of age — A total of 30 subjects will perform four tasks per person for a single task (motor task) and a double task (motor task + cognitive task), and the test order will be randomly assigned. The subject's prefrontal cortex activity will be measured using fNIRS (NIRSIT, OBELAB).
  The single task will be to perform a 10-meter walk test and an 8-way walk test as exercise tasks. as not affected by acceleration and deceleration. The dual task will be carried out together with the exercise task and the cognitive task. The cognitive task will be a simple calculation problem so that it can be performed without much difficulty when walking.Subjects will perform a total of three iterations and have a break of 20 seconds before each task begins.

SUMMARY:
The goal of this observational study is to compare to investigate the effect of dual task performance on straight and curved walking in elderly people with mild cognitive impairment.

The main question[s] it aims to answer are:

* The purpose of this study was to investigate the effect of dual task performance on the activity of the prefrontal cortex in the elderly with mild cognitive impairment during straight and curved walking.
* The purpose of this study was to investigate the effect of dual task performance on gait speed during straight and curved walking in elderly people with mild cognitive impairment.

Participants will: For mild cognitive impairment 65 and older who can do dual tasks.

* single task (motor task) : an exercise task, which will perform a 10-meter walking test and a figure-eight walking test.
* double task (motor task + cognitive task) : planned to perform a motor task and a cognitive task together. The cognitive task is scheduled to be a simple calculation problem so that it can be performed without great difficulty while walking.

DETAILED DESCRIPTION:
The goal of this observational study is to compare to investigate the effect of dual task performance on straight and curved walking in elderly people with mild cognitive impairment.

The main question[s] it aims to answer are:

* The purpose of this study was to investigate the effect of dual task performance on the activity of the prefrontal cortex in the elderly with mild cognitive impairment during straight and curved walking.
* The purpose of this study was to investigate the effect of dual task performance on gait speed during straight and curved walking in elderly people with mild cognitive impairment.

Participants will A total of 30 subjects will perform a single task (motor task) and a double task (motor task + cognitive task), four tasks per subject, and the order of examination will be randomly assigned. The subject's prefrontal cortex activity will be measured using fNIRS (NIRSIT, OBELAB).

The single task is an exercise task, which will perform a 10-meter walking test and a figure-eight walking test. The 10-meter walking test was developed to evaluate walking speed during short distance walking.

The total length was set to 14 m, and a distance of 2 m was placed at the beginning and end to avoid being affected by acceleration and deceleration. The figure-eight gait test requires a person to walk in a figure-eight shape around two cones placed as a tool to measure curved walking ability. In this study, in order to perform the exercise task at the same distance, a straight line of 14 m will be made into a random line and set in the shape of a figure 8.

Do not deviate more than 1 m from the object in the rotating section of the object. The dual task is planned to perform a motor task and a cognitive task together. The cognitive task is scheduled to be a simple calculation problem so that it can be performed without great difficulty while walking. The subject will perform a total of 3 repetitions and will have a 20-second break before starting each task.

ELIGIBILITY:
Inclusion Criteria:

* A person with a Korean version of the Simplified Mental Status Test (K-MMSE-2) score of 18-23.
* A person who can walk using an auxiliary device.

Exclusion Criteria:

* A person who cannot walk 3 meters back and forth or stand up from a sitting position
* A person sensitive to infrared lasers
* A person with impaired vision and hearing

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: For mild cognitive impairment 65 and older who can do dual tasks.
Sampling Method: Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2023-05-31 (Actual); Primary Completion 2023-06-05 (Actual); Study Completion 2023-06-05 (Actual)

PRIMARY OUTCOMES:
prefrontal cortex activity for single and dual tasks | through study completion, an average of 1 week.
  functional near-infrared spectroscopy : fNIRS, a non-invasive vascular-based neuroimaging technology, is a tool that uses light sources and photoreceptors to measure changes in the concentration of oxyhemoglobin (HbO2) in the cerebral cortex area due to the regulation of neural activity.
  In this study, fNIRS measurements were performed by a wireless cw system (NIRSIT, OBELAB, Republic of Korea) an fNIRS device consisting of five double wavelength (780/850 nm) laser sources and seven detectors. The amount of HbO₂ change while performing the task were measured. The device consists of 15 channels with a distance of 30 mm between each pair.
Walking speed for single and dual tasks | through study completion, an average of 1 week.
  Using a stopwatch, real-time measurements will be made in the remaining sections except for the front and back 2m, considering acceleration and deceleration when walking along a straight 14m path and a curved path.

CONTACTS AND LOCATIONS:
Overall Officials: YuMin Lee, MS candidate, Principal Investigator — Sahmyook University
Locations (1):
- Sahmyook university, Seoul, Nowon-gu, South Korea